CLINICAL TRIAL: NCT04725903
Title: Extended-Field Lymph Node Proton Irradiation for High Risk Prostate Cancer
Brief Title: Proton Radiation Therapy for the Treatment of Patients with High Risk Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Pretesh Patel, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000329; NCI-2020-07113 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RAD5131-20 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2021-01-08; First posted 2021-01-27 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Stage III Prostate Cancer AJCC V8; Stage IIIA Prostate Cancer AJCC V8; Stage IIIB Prostate Cancer AJCC V8; Stage IIIC Prostate Cancer AJCC V8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy; Proton Therapy; Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (proton beam therapy) (Experimental): Patients undergo conventionally fractionated or hypofractionated proton beam therapy daily on Monday-Friday directed to the prostate, pelvic lymph nodes, and para-aortic lymph nodes. Patients may receive an optional high-dose rate brachytherapy boost. Androgen deprivation therapy is required but left to the discretion of the treating physician.
  Interventions: Radiation: High-Dose Rate Brachytherapy; Radiation: Proton Beam Radiation Therapy; Other: Quality-of-Life Assessment; Other: Survey Administration

INTERVENTIONS:
Radiation: High-Dose Rate Brachytherapy — Receive high-dose rate brachytherapy boost
  Other Names: Brachytherapy, High Dose
Radiation: Proton Beam Radiation Therapy — Undergo proton beam therapy
  Other Names: PBRT; Proton; Proton Radiation Therapy; Radiation, Proton Beam
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Survey Administration — Ancillary studies

SUMMARY:
This phase II trial investigates whether proton radiation therapy directed to the prostate tumor, pelvic, and para-aortic lymph nodes, is an effective way to treat patients with high-risk or lymph node positive prostate cancer who are receiving radiation therapy, and if it will result in fewer gastrointestinal and genitourinary side effects. Proton beam therapy is a new type of radiotherapy that directs multiple beams of protons (positively charged subatomic particles) at the tumor target, where they deposit the bulk of their energy with essentially no residual radiation beyond the tumor. By reducing the exposure of the healthy tissues and organs to radiation in the treatment of prostate cancer, proton therapy has the potential to better spare healthy tissue and reduce the side effects of radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the rate of acute grade 2+ gastrointestinal toxicity compared to historical photon treatments.

SECONDARY OBJECTIVES:

I. To determine the rate of acute grade 2+ genitourinary toxicity compared to historical photon treatments.

II. To assess the feasibility of extended-field proton irradiation of high-risk prostate.

III. To demonstrate safety of proton therapy followed by high dose rate (HDR) boost.

IV. To determine patient-reported outcomes (PROs) of toxicity.

OUTLINE:

Patients undergo conventionally fractionated proton beam therapy daily on Monday-Friday. Patients may receive a high-dose rate brachytherapy boost.

After completion of study treatment, patients are followed up at 1, 3, 6, 9 and 12 months, and 1.5, 2, 2.5, and 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed high-risk prostate cancer fulfilling any one of the following criteria:

  * Gleason grade 8 or higher
  * cT3b (seminal vesicle involvement) or cT4
  * Prostate specific antigen [PSA] > 20 (or PSA >10 if on finasteride)
  * Clinically or pathologically positive regional lymph nodes within the inguinal, external iliac, internal iliac, obturator, peri-rectal, pre-sacral, common iliac, or lower para-oaortc (inferior to the L2-L3 interspace) basins
* Zubrod performance status 0-2
* Complete blood cell (CBC)/differential obtained within 90 days prior to registration on study
* Absolute neutrophil count (ANC) >= 1,500 cells/mm^3
* Platelets >= 100,000 cells/mm^3
* Hemoglobin >= 8.0 g/dl (Note: The use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 8.0 g/dl is acceptable)
* Patient must be able to provide study specific informed consent

Exclusion Criteria:

* Absence of bone metastasis by bone scan or metabolic imaging (e.g. NaF PET, FACBC PET, PSMA PET, etc.) before the start of therapy.
* Absence of distant lymph node metastasis by CT and/or MRI before the start of therapy.
* Previous radical surgery (prostatectomy) or cryosurgery for prostate cancer
* Prior radiotherapy, including brachytherapy, to the region of the study cancer that would result in overlap of radiation therapy fields
* Uncontrolled intercurrent illness including, but not limited to, inflammatory bowel disease, human immunodeficiency virus infection, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute grade 2+ gastrointestinal (GI) toxicity | Up to 3 years
  The rate of grade 2+ gastrointestinal toxicity within 30 days of receiving radiation therapy (RT) will be measured. It will be compared to the theorized reduction to 24% toxicity using the exact binomial test. Assessments are based on version 5 Common Terminology Criteria for Adverse Events (CTCAE), and the worst severity of GI toxicity will be assessed.

SECONDARY OUTCOMES:
Acute grade 2+ genitourinary (GU) toxicity rate | Up to 3 years
  The rate of grade 2+ genitourinary toxicity within 30 days of receiving radiation therapy (RT) will be measured. Assessments are based on version 5 CTCAE, and the worst severity of GU toxicity will also be assessed.
Optimal frequency of cone beam computed tomography (CT) | Through study completion, an average of 1 year
  Will determine the optimal frequency of cone beam CT during treatment and assess subsequent need for adaptive re-planning. The feasibility of extended-field proton irradiation of high-risk prostate cancer will be estimated using a re-planning rate of less than 10%. The re-planning rate will be estimated as binary variable, yes or no. The exact 95% confidence interval (CI) around the 10 % re-planning count based on the binomial distribution for the estimated 30 patients will be used (0.021-0.265). The study will be deemed feasible if the observed rate is not higher than the upper bound of the estimated 95% CI.
Patient reported health related quality of life (QOL) - PRO-CTCAU GI | Up to 3 years
  Assessed using Patient Reported Outcomes-CTCAE GI toxicity
Patient reported health related quality of life (QOL) - PRO-CTCAU GU | Up to 3 years
  Assessed using Patient Reported Outcomes-CTCAE GU toxicity
Patient reported health related quality of life (QOL) - IPSS | Up to 3 years
  International Prostate Symptom Score (IPSS)
Patient reported health related quality of life (QOL) - EPIC-CP | Up to 3 years
  Expanded Prostate Cancer Index Composite for Clinical Practice (EPIC-CP)
Chronic GI Toxicity | Up to 3 years
  The rate of any grade gastrointestinal toxicity occurring after 90 days from the completion of radiation therapy(RT). Assessments are based on version 5 Common Terminology Criteria for Adverse Events (CTCAE), and the worst severity of GI toxicity will be assessed.
Chronic GU Toxicity | Up to 3 years
  The rate of any grade genitourinary toxicity occurring after 90 days from the completion of radiation therapy(RT). Assessments are based on version 5 Common Terminology Criteria for Adverse Events (CTCAE), and the worst severity of GU toxicity will be assessed.
Biochemical failure | Baseline up to pre-RT
  Assessed by the Phoenix definition (prostate specific antigen [PSA] >= 2 ng/ml over the nadir PSA).

CONTACTS AND LOCATIONS:
Overall Officials: Pretesh R Patel, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
Results of the trial and not individual patient data will be shared. The study protocol, consent, and investigator's brochure will be available. The statistical plan is incorporated into the protocol, along with inclusion and exclusion criteria.